CLINICAL TRIAL: NCT02289599
Title: A Randomized, Double-blind, Placebo-controlled, Single-Ascending Dose Study to Assess Safety, Tolerability, and Pharmacokinetics of E2307 in Healthy Young and Elderly Japanese Subjects
Brief Title: A Study to Assess Safety, Tolerability, and Pharmacokinetics of E2307 in Healthy Young and Elderly Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2307-J081-001
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Healthy Subjects
Keywords: Healthy Japanese Subjects; E2307; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Part A: 1 mg E2307 (young cohort) (Experimental): E2307 (1 x 1 mg E2307 capsule) or placebo (1 x 1 E2307 matching placebo capsule)
  Interventions: Drug: E2307; Drug: E2307 Matching Placebo
- Part A: 3 mg E2307 (young cohort) (Experimental): E2307 (3 x 1 mg E2307 capsules) or placebo (3 x 1 E2307 matching placebo capsules)
  Interventions: Drug: E2307; Drug: E2307 Matching Placebo
- Part A: 10 mg E2307 (young cohort) (Experimental): E2307 (1 x 10 mg E2307 capsule) or placebo (1 x 1 E2307 matching placebo capsule)
  Interventions: Drug: E2307; Drug: E2307 Matching Placebo
- Part A: 30 mg E2307 (young cohort) (Experimental): E2307 (3 x 10 mg E2307 capsules) or placebo (3 x 1 E2307 matching placebo capsules)
  Interventions: Drug: E2307; Drug: E2307 Matching Placebo
- Part A: 100 mg E2307 (young cohort) (Experimental): E2307 (1 x 100 mg E2307 capsule) or placebo (1 x 1 E2307 matching placebo capsule)
  Interventions: Drug: E2307; Drug: E2307 Matching Placebo
- Part A: 200 mg E2307 (young cohort) (Experimental): E2307 (2 x 100 mg E2307 capsules) or placebo (2 x 1 E2307 matching placebo capsules)
  Interventions: Drug: E2307; Drug: E2307 Matching Placebo
- Part A: 300 mg E2307 (young cohort) (Experimental): E2307 (3 x 100 mg E2307 capsules) or placebo (3 x 1 E2307 matching placebo capsules)
  Interventions: Drug: E2307; Drug: E2307 Matching Placebo
- Part B: Elderly cohort (Experimental): One dose level below MTD from Part A
  Interventions: Drug: E2307

INTERVENTIONS:
Drug: E2307
Drug: E2307 Matching Placebo
  Arms: Part A: 1 mg E2307 (young cohort); Part A: 10 mg E2307 (young cohort); Part A: 100 mg E2307 (young cohort); Part A: 200 mg E2307 (young cohort); Part A: 3 mg E2307 (young cohort); Part A: 30 mg E2307 (young cohort); Part A: 300 mg E2307 (young cohort)

SUMMARY:
This study will be a single-center, single dose, randomized, double-blind, placebo-controlled study in healthy Japanese male subjects. The study will consist of 2 parts: Part A (young subjects) and Part B (elderly subjects). In Part A sequential cohorts of subjects will be treated with single ascending doses of E2307. The maximum tolerated dose (MTD) will be determined in Part A. Part B will be initiated after Part A is completed. In Part B one cohort of healthy elderly subjects will be treated with a single dose of E2307 at one dose level below the MTD. In part A, a total of 56 subjects will be enrolled into 7 cohorts sequentially and randomized 3:1 to receive either E2307 (1 mg, 3 mg, 10 mg, 30 mg, 100 mg, 200 mg, or 300 mg) or placebo. In part B, a total of 8 subjects will be randomized, 6 subjects to a single dose of E2307 and 2 subjects to placebo.

ELIGIBILITY:
Inclusion Criteria:

Parts A and B

1. Provide written informed consent
2. Willing and able to comply with all aspects of the protocol

   Part A: Young cohort
3. Non-smoking, male subjects age >=20 years and less than 55 years old at the time of informed consent

   Part B: Elderly Cohort
4. Non-smoking, male subjects age >=65 years and less than 85 years old at the time of informed consent

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from this study:

1. Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks of dosing
2. Any history of abdominal surgery that may affect PK profiles of E2307 (eg. hepatectomy, nephrectomy, digestive organ resection)
3. Known history of clinically significant drug allergy (at Screening)

Ages: 20 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-11; Primary Completion 2015-02 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Number of adverse events/serious adverse events | Up to 30 days
Plasma pharmacokinetics (PK) of E2307: Cmax (maximum observed concentration) | Up to 12 days
Plasma PK of E2307: tmax (time at which the highest drug concentration occurs) | Up to 12 days
Plasma PK of E2307: AUC(0-t) [area under the concentration (AUC)-time curve from zero time to time of last quantifiable concentration] | Up to 12 days
Plasma PK of E2307: AUC(0-inf) [area under the concentration-time curve from zero time extrapolated to infinite time] | Up to 12 days
Plasma PK of E2307: t1/2 (terminal elimination phase half-life) | Up to 12 days
Plasma PK of E2307: CL/F (apparent total clearance following oral administration) | Up to 12 days
  CL/F are calculated for E2307 only
Plasma PK of E2307: Vz/F (apparent volume of distribution at terminal phase) | Up to 12 days
  Vz/F are calculated for E2307 only
Plasma PK of E2307: AUC ratio (AUC ratio of metabolite to parent) | Up to 12 days
Urine PK of E2307: Ae (cumulative amount of drug excreted in urine up to 264 hours postdose) | Up to 12 days
Urine PK of E2307: CLR (renal clearance) | Up to 12 days

SECONDARY OUTCOMES:
Mean difference in change of mean blood pressure (BP) between E2307 and placebo | 24 hours predose and continue until 24 hours postdose (Day 2)
QT interval assessment using Holter monitoring | 24 hours predose through Day 2 (at 24 hours postdose)

CONTACTS AND LOCATIONS:
Locations (1):
- Kagoshima, Kagoshima-ken, Japan